CLINICAL TRIAL: NCT04950738
Title: The Effectiveness of Acupuncture for Complications in Critically Ill Patients: Multiple Centers a Double-Blind Randomized Control Trial
Brief Title: The Effectiveness of Acupuncture for Complications in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, Principal Investigator, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CMUH110-REC1-037
Record Dates: First submitted 2021-06-22; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Delirium; Agitation; Arrhythmia; Feeding Intolerance; Pain, Acute
Keywords: acupuncture; intensive care; delirium; agitation; double blinded randomized control study
MeSH Terms: conditions — Delirium; Psychomotor Agitation; Arrhythmias, Cardiac; Acute Pain

STUDY DESIGN:
Intervention Model Description: multicenter parallel arm double-blind randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture with press tack needle group (Acu) (Experimental): Patients in acupuncture group will receive traditional Chinese acupuncture using Press Tack Needle (PYONEX 0.20 x l.5mm made by Seirin Corporation). The following acupoints will be used: HT 7 (Shen Men), PC 6 (Nei Guan), LU 9 (Tai yuan), LI 4 (He Gu), SP 3 (Tai Bai,) ST 44 (Nei ting), LIV 3 (Tai Chong). The treatment will use bilateral acupuncture Interventions will be given on day 1, 3, and 5 after patient's enrolment.
  Interventions: Other: pess tack acupuncture
- Placebo group press tack placebo (Con) (Placebo Comparator): Patients randomized to the control group will receive a press lack placebo (made by Seirin Corporation), which looks identical to press tack needles but, with no needle element. The point selection will be identical to the acupuncture group: HT 7 (Shen Men), PC 6 (Nei Guan), LU 9 (Tai yuan), L1 4 (He Gu), SP 3; (Tat Bai), ST 44 (Ne1 tmg), LIV 3 (Tat Chong). Interventions will be given on days 1, 3, and 5 after the patient's enrolment.
  Interventions: Other: pess tack placebo

INTERVENTIONS:
Other: pess tack acupuncture — Patients enrolled will receive intervention in a form of either press tack acupuncture needles or press tack placebos. Three total intervention sessions will be taken place on day 1,3,5 from patient's enrolment. Needles/placebos skin withdrawal will be done 48 hours after treatment by an acupuncture doctor or by a trained ICU nurne. In cases when a patient will be transferred from the ICU, the 3 study interventions will be continued in the new ward.
  Other Names: Press Tack Needle/ sticker needle/ PYONEX
  Arms: Acupuncture with press tack needle group (Acu)
Other: pess tack placebo — pess tack stickers without a needle
  Other Names: PYONEX placebo
  Arms: Placebo group press tack placebo (Con)

SUMMARY:
Introduction:

Intensive care unit (ICU) is a special department in the health care facility. Although with high development of modern medicine nowadays, the average mortality rate in ICU is still around 7 to 20 %. There are a few tricky problems that intensivists and ICU nurses faced very often, including ICU delirium, arrhythmia and poor digestion problem that will all affect the mortality and morbidity rate of critical care patients.

Methods: A randomized control trial will examine the effect of press tack acupuncture vs. press tack placebos. The patients will be randomly divided (1:1) into one of two groups. A total of 80 ICU patients will have to meet the following criteria: age 20-90, newly ICU admission(<48 hours), APACHE score <30, one or no inotropic medicine use, FiO2< 60%. Three interventions will be given in each group. The main outcomes will be the incidence of arrhythmia, delirium, and poor digestion and the severity of pain. We will also record ICU mortality, ICU stays and hospital days.

DETAILED DESCRIPTION:
Introduction:

Intensive care unit (ICU) is a special department in the health care facility. Although with high development of modern medicine nowadays, the average mortality rate in ICU is still around 7 to 20 %. There are a few tricky problems that intensivists and ICU nurses faced very often, including ICU delirium, arrhythmia and poor digestion problem that will all affect the mortality and morbidity rate of critical care patients.

Methods: A randomized control trial will examine the effect of press tack acupuncture vs. press tack placebos. The patients will be randomly divided (1:1) into one of two groups. A total of 80 ICU patients will have to meet the following criteria: age 20-90, newly ICU admission(<48 hours), APACHE score <30, one or no inotropic medicine use, FiO2< 60%. Three interventions will be given in each group. The main outcomes will be the incidence of arrhythmia, delirium, and poor digestion and the severity of pain. We will also record ICU mortality, ICU stays and hospital days.

Expected outcome: The study finding will help to determine the therapeutic effect of acupuncture for ICU complications.

Other information: This study will be conducted in the ICU departments of China medical hospital and Asia University Hospital, Taichung city, Taiwan. The study is conducted on stable ICU patients and we don't anticipate any serious risk for adverse events following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 20--90

  * newly ICU admission (<48 hours)
  * APACHE score <30
  * Less than 3 inotropic medicine use
  * Fi02< 60%.

Exclusion Criteria:

* • Coagulopathy: Prolong Prothrombin Time (PPT) activated Partial Thromboplastin Time (aPTT) more than 4 times

  * Thrombocytopenia - low platelet count
  * Clinically unstable: receiving two or more inotropic agents or Fraction of Inspired Oxygen (Fi02) >60%
  * Primary central nervous system disorder: stroke, traumatic brain injury, central nervous system infections, brain tumors, recent intracranial surgery
  * Already under other traditional medicine intervention during hospitalization
  * Skin damage of more than 20% of the body skin.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
arrhythmia | at the patient's ICU discharge, on average 1 week
  incidence of arrhythmia
delirium | at the patient's ICU discharge, on average 1 week
  4 or more points according to the Intensive Care Delirium Screening Checklist (ICDSC)(0-8 scale, score of less than 4 points indicate no delirium, 4 or more indicate delirium) and a Richmond Agitation-Sedation Scale (RASS) score of: +l, +2, +3, +4 - 1, -2 (score meanings +1 - 4 = levels of agitation, -1-4= levels of sudation, 0 = normal mental state.
feeding intolorance | at the patient's ICU discharge, on average 1 week
  measured by days to reach the target Energy Fxpenditure
pain in the intensive care unit (ICU) | at the patient's ICU discharge, on average 1 week
  For pain the Numeric Rating scale will be applied in patients that are able to express their self. As well as the Behavioral pain scale. The Critical Care Pain Observation Tool (CPOT) 0-8, will also be filled by the doctor and nurses along with the dose of fentanyl, hydromorphone methadone, morphine, and remifentanil and other analgesic medications.
dose of arrhythmia drugs | at the patient's ICU discharge, on average 1 week
  the dose of Adenosine, calcium channel blockers, or beta-blocking agents or other arrhythmia drugs
  .
dose of use of prokinetic drugs | at the patient's ICU discharge, on average 1 week
  does of metoclopramide, Erythromycin or other prokinetic drugs
analgesic medication use | at the patient's ICU discharge, on average 1 week
  dose of fentanyl, hydromorphone methadone, morphine, and remifentanil and other analgesic medications.
delirium drug use | at the patient's ICU discharge, on average 1 week
  addition to drug use (a daily dose of sedative drugs, muscle relaxant, or atypical antipsychotics IV Haloperidol Benzodiazepines, Precedex, Propofol and oral Quediapine)

SECONDARY OUTCOMES:
the use of Parental nutrition | at the patient's ICU discharge, on average 1 week
  patients who cannot digest with daily NG tube: drainage: more than 500ml per day or severe diarrhea more the 1000 ml per day
the need for a post-pyloric tube | at the patient's ICU discharge, on average 1 week
  patients who cannot digest with daily NG tube and by doctor decision
vomitus | at the patient's ICU discharge, on average 1 week
  in microliters
diarrhea | at the patient's ICU discharge, on average 1 week
  in microliters
constipation days | at the patient's ICU discharge, on average 1 week
  3 days without stool discharge
gastrointestinal (GI) bleeding | at the patient's ICU discharge, on average 1 week
  in number of times
albumin blood levels | at the patient's ICU discharge, on average 1 week
  serum albumin blood levels
Intravenous (IV) injected albumin | at the patient's ICU discharge, on average 1 week
  IV injected albumin in grams
heart rate | day 1,3,5,7
  number of beats per minute
blood pressure | day 1,3,5,7
  systolic and diastolic blood pressure in mm Hg
SpO2 oxygen saturation | day 1,3,5,7
  Sp02 oxygen saturation levels
Respiratory rate | day 1,3,5,7
  measured by number of breath in one minute
mean arterial pressure | day 1,3,5,7
  average pressure in a patient's arteries during one cardiac cycle
Body temperature | at the patient's ICU discharge, on average 1 week
  number of days of body temperature over 38 °C
ventilator data | day 1,3,5,7
  ventilator data
Overall Satisfaction of patient family | at the patient Hospital discharge, on average 1 month
  Overall Satisfaction of patient family will be measured by the European Family Satisfaction with Care in the Intensive Care Unit (EURO FS-ICU).
mechanical ventilation days days | at the patient Hospital discharge, on average 1 month
  number of days under mechanical ventilation
ICU stay | at the patient's ICU discharge, on average 1 week
  number of admission days to the ICU
hospital days | at the patient Hospital discharge, on average 1 month
  number of admission days to the hospital
ICU mortality | at the patient's ICU discharge, on average 1 week
  number of patients died in the ICU
Hospital mortality | at the patient Hospital discharge, on average 1 month
  number of patients died in the hospital
cost of hospital admission | at the patient Hospital discharge, on average 1 month
  cost of hospital admission in New Taiwan Dollars {TWD)
cost of ICU admission | at the patient's ICU discharge, on average 1 week
  cost of ICU admission in New Taiwan Dollars {TWD).
acupuncturist blinding | after intervention on day 5
  blinding questioner will ask the acupuncturist to which group he/she guessed he/she applied the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chen Lee, Principal Investigator — China Medical University Hospital

IPD SHARING:
Plan to Share IPD: No